CLINICAL TRIAL: NCT04938323
Title: Prevention of Acute Respiratory Infection in Taiwanese Institutionalized Elderly (PARITIE)
Brief Title: Prevention of Acute Respiratory Infection in Taiwanese Institutionalized Elderly
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Covid-19 related delays in project launch
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: Chang-Hua Hospital (Other Government)
Responsible Party: Principal Investigator, Megan Murray, MD, ScD, Professor of Global Health, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB20-0661
Record Dates: First submitted 2021-05-28; First posted 2021-06-24 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Acute Respiratory Infection
MeSH Terms: interventions — BCG Vaccine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 allocation to receive intradermal administration of BCG vaccination or placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and investigators will be blinded. Designated staff whose responsibility will be to administer the BCG vaccine or placebo will not be blinded. These designated staff members will not be involved in the collection of outcome data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCG Vaccine (Experimental): Participants randomized to the BCG Vaccine Arm will receive the vaccine. The vaccination site is about halfway down the outer aspect of the upper arm.
  Interventions: Drug: BCG Vaccine
- Placebo Arm (Placebo Comparator): Placebo will be administered in an intradermal route in the same location as the BCG vaccines': upper arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BCG Vaccine — .1 mL of reconstituted BCG vaccine given intradermally at baseline.
  Arms: BCG Vaccine
Drug: Placebo — .1 mL of diluent (saline) given intradermally at baseline
  Arms: Placebo Arm

SUMMARY:
The purpose of this study is to assess the efficacy of Bacille Calmette-Guérin (BCG) vaccination compared to placebo against acute respiratory infections in the elderly who are less protected by standard vaccines against influenza than other age groups. The investigators hypothesize that BCG vaccination can reduce incidence of infection and severity of a range of acute respiratory infections. Patients who are residents of participating long-term care facilities (LTCFs), who agree to participate in the study, or with a legal guardian who agrees on their behalf, will be randomly assigned to receive BCG vaccination or a placebo. Participants will be followed for up to six months to assess the incidence of infection and the severity of a range of acute respiratory infections.

DETAILED DESCRIPTION:
This is a Phase III, double-blind, randomized placebo-controlled trial comparing efficacy of BCG vaccination to that of placebo in reducing severity of a range of acute respiratory infections. Participants will need to meet eligibility criteria in order to be included in the study. Those selected will be asked to provide a blood sample for complete blood count, liver function and renal tests, tests to calculate MELD score, also serological testing.

Participants will be randomized in a 1:1 allocation to receive intradermal administration of BCG vaccination or placebo at baseline. During follow-up, the study team will monitor participants' health status by using intermittent surveys about the presence of adverse events potentially related to vaccination, clinic visits or hospitalization for acute respiratory infection, BioFire® Respiratory 2.1 panel for respiratory pathogens and disease outcome status.

The investigators will screen 980 individuals to enroll 830 participants, resulting in 415 receiving BCG vaccine and 415 receiving placebo. The proposed enrollment sample size is designed to provide 80% power to detect 60% vaccine efficacy (a relative risk of 0.4 among the vaccinated) with 0.05 type-1 error in a two-tailed test, assuming 10% lost to follow-up. The number of individuals screened assumes about 15% will not be eligible to be enrolled after screening.

Objective: To measure the impact of one-time BCG-Japan vaccination on acute respiratory infections leading to hospitalization in the elderly.

Primary Endpoint 1: The cumulative incidence of hospitalization for acute respiratory infection following BCG vaccination compared to that following placebo, starting from 14 days post-vaccination, as defined using relevant ICD-10 codes.

If BCG vaccine is shown to be effective in this age group, it will be of major benefit to both study participants and other elderly individuals at risk for acute respiratory infections and have added protection from disease. Identification of an intervention that can reduce the risk of infection and/or of being hospitalized with ARI would reduce the number of new cases and reducing the number of cases that require hospital admission and vast resources.

ELIGIBILITY:
Inclusion Criteria:

* Clients of a long-term care facility
* 55-85 years old

Exclusion Criteria:

* Known previous or current active TB disease
* Exposure to individual with documented active TB within previous three months
* Fever (>37.5 C) within the past 24 hours
* Current serious underlying medical conditions:

  * HIV+
  * Currently taking immunosuppressive or immunomodulatory drugs
  * Expect to receive chemotherapy or radiation therapy in the coming six months, receipt of chemotherapy in the past six months or undergoing chemotherapy
  * Currently on any anti-cytokine therapy
  * History of organ or bone marrow transplantation
  * Individual or family history of familial or acquired immune disorder, including auto-immune disorders
  * Neutropenia/leukopenia (<500 neutrophils/mm3 or <400 lymphocytes/mm3)
  * Chronic kidney disease (Glomerular Filtration Rate< 30 ml/min/1.73m2)
  * Elevated liver enzymes (alanine aminotransferase >260 IU/L or aspartate aminotransferase >200 IU/L) or Model for End-Stage Liver Disease (MELD) score ≥30
  * Treatment with oral or intravenous steroids at the time of screening, defined as daily doses of 10mg prednisone or equivalent for longer than 3 months.
  * Solid or hematologic malignancy including lymphoma, leukemia and other reticuloendothelial system carcinomas within the past two years.
  * Presence of Parkinson's disease
  * Evidence of dermatitis at site of vaccination
* Living with someone with HIV, immunocompromised, taking immunosuppressive drugs
* Suspicion of active viral or bacterial infection, or taking antivirals or antibiotics
* Any vaccine administration two weeks before or after BCG administration. For those who have received the Covid-19 vaccine, the two weeks are considered after the 2nd dose.

  * Doctors in Taiwan do not always encourage the use of Covid-19 vaccination due to low incidence of disease and the risk of death due to blood clots in the only approved vaccine for use (AstraZeneca).
* Known allergy to components of the BCG vaccine or prior serious reaction to previous BCG administration
* Plan to leave the long-term care facility within the next three months
* Taking part in any ongoing trial that includes administration of an investigational product relevant to respiratory disease
* Participants with cognitive impairment whose legal guardians cannot be contacted

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
To measure the impact of one-time BCG vaccination compared to placebo in reducing the occurrence of acute respiratory infection leading to hospitalization in the elderly in Taiwan | 6 months
  Number of hospitalizations for acute respiratory infection as defined by list of ICD codes

SECONDARY OUTCOMES:
To measure the impact of one-time BCG vaccination compared to placebo in reducing the occurrence of medically attended acute respiratory infection | 6 months
  Number of medically attended acute respiratory infection
To measure the impact of one-time BCG vaccination compared to placebo on microbiologically confirmed viral respiratory illness | 6 months
  Number of microbiologically confirmed viral respiratory illness by viral pathogen as measure by BioFire® Respiratory 2.1 PCR panel
To measure the impact of one-time BCG vaccination compared to placebo on duration of hospitalization due to acute respiratory infection during the study follow-up period | 6 months
  Total duration of days spent hospitalized due to acute respiratory infection during the study follow-up period
To measure the impact of one-time BCG vaccination compared to placebo on critical admissions during the follow-up period | 6 months
  Number of critical are admissions during the follow-up period
To measure the impact of one-time BCG vaccination compared to placebo on all-cause mortality deaths | 6 months
  Number of all-cause mortality deaths
To measure the impact of one-time BCG vaccination compared to placebo on local and systemic adverse events | 6 months
  Number of local and systemic adverse events to BCG vaccination following randomization
To measure the impact of one-time BCG vaccination compared to placebo on changes of antibody profiles | 6 months
  Number of changes in antibody profiles between enrollment and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Megan Murray, ScD, Principal Investigator — Harvard Medical School (HMS and HSDM)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ritz N, Hanekom WA, Robins-Browne R, Britton WJ, Curtis N. Influence of BCG vaccine strain on the immune response and protection against tuberculosis. FEMS Microbiol Rev. 2008 Aug;32(5):821-41. doi: 10.1111/j.1574-6976.2008.00118.x. Epub 2008 Jul 9. PMID 18616602
- [Background] Abubakar I, Pimpin L, Ariti C, Beynon R, Mangtani P, Sterne JA, Fine PE, Smith PG, Lipman M, Elliman D, Watson JM, Drumright LN, Whiting PF, Vynnycky E, Rodrigues LC. Systematic review and meta-analysis of the current evidence on the duration of protection by bacillus Calmette-Guerin vaccination against tuberculosis. Health Technol Assess. 2013 Sep;17(37):1-372, v-vi. doi: 10.3310/hta17370. PMID 24021245
- [Background] Walk J, de Bree LCJ, Graumans W, Stoter R, van Gemert GJ, van de Vegte-Bolmer M, Teelen K, Hermsen CC, Arts RJW, Behet MC, Keramati F, Moorlag SJCFM, Yang ASP, van Crevel R, Aaby P, de Mast Q, van der Ven AJAM, Stabell Benn C, Netea MG, Sauerwein RW. Outcomes of controlled human malaria infection after BCG vaccination. Nat Commun. 2019 Feb 20;10(1):874. doi: 10.1038/s41467-019-08659-3. PMID 30787276
- [Background] Koeken VACM, Verrall AJ, Netea MG, Hill PC, van Crevel R. Trained innate immunity and resistance to Mycobacterium tuberculosis infection. Clin Microbiol Infect. 2019 Dec;25(12):1468-1472. doi: 10.1016/j.cmi.2019.02.015. Epub 2019 Feb 23. PMID 30807849
- [Background] Suliman S, Geldenhuys H, Johnson JL, Hughes JE, Smit E, Murphy M, Toefy A, Lerumo L, Hopley C, Pienaar B, Chheng P, Nemes E, Hoft DF, Hanekom WA, Boom WH, Hatherill M, Scriba TJ. Bacillus Calmette-Guerin (BCG) Revaccination of Adults with Latent Mycobacterium tuberculosis Infection Induces Long-Lived BCG-Reactive NK Cell Responses. J Immunol. 2016 Aug 15;197(4):1100-1110. doi: 10.4049/jimmunol.1501996. Epub 2016 Jul 13. PMID 27412415
- [Background] Nemes E, Geldenhuys H, Rozot V, Rutkowski KT, Ratangee F, Bilek N, Mabwe S, Makhethe L, Erasmus M, Toefy A, Mulenga H, Hanekom WA, Self SG, Bekker LG, Ryall R, Gurunathan S, DiazGranados CA, Andersen P, Kromann I, Evans T, Ellis RD, Landry B, Hokey DA, Hopkins R, Ginsberg AM, Scriba TJ, Hatherill M; C-040-404 Study Team. Prevention of M. tuberculosis Infection with H4:IC31 Vaccine or BCG Revaccination. N Engl J Med. 2018 Jul 12;379(2):138-149. doi: 10.1056/NEJMoa1714021. PMID 29996082
- [Background] Kleinnijenhuis J, Quintin J, Preijers F, Joosten LA, Ifrim DC, Saeed S, Jacobs C, van Loenhout J, de Jong D, Stunnenberg HG, Xavier RJ, van der Meer JW, van Crevel R, Netea MG. Bacille Calmette-Guerin induces NOD2-dependent nonspecific protection from reinfection via epigenetic reprogramming of monocytes. Proc Natl Acad Sci U S A. 2012 Oct 23;109(43):17537-42. doi: 10.1073/pnas.1202870109. Epub 2012 Sep 17. PMID 22988082
- [Background] Spencer JC, Ganguly R, Waldman RH. Nonspecific protection of mice against influenza virus infection by local or systemic immunization with Bacille Calmette-Guerin. J Infect Dis. 1977 Aug;136(2):171-5. doi: 10.1093/infdis/136.2.171. PMID 894076
- [Background] Netea MG, Joosten LA, Latz E, Mills KH, Natoli G, Stunnenberg HG, O'Neill LA, Xavier RJ. Trained immunity: A program of innate immune memory in health and disease. Science. 2016 Apr 22;352(6284):aaf1098. doi: 10.1126/science.aaf1098. Epub 2016 Apr 21. PMID 27102489
- [Background] Arts RJW, Moorlag SJCFM, Novakovic B, Li Y, Wang SY, Oosting M, Kumar V, Xavier RJ, Wijmenga C, Joosten LAB, Reusken CBEM, Benn CS, Aaby P, Koopmans MP, Stunnenberg HG, van Crevel R, Netea MG. BCG Vaccination Protects against Experimental Viral Infection in Humans through the Induction of Cytokines Associated with Trained Immunity. Cell Host Microbe. 2018 Jan 10;23(1):89-100.e5. doi: 10.1016/j.chom.2017.12.010. PMID 29324233
- [Background] Netea MG, van Crevel R. BCG-induced protection: effects on innate immune memory. Semin Immunol. 2014 Dec;26(6):512-7. doi: 10.1016/j.smim.2014.09.006. Epub 2014 Oct 23. PMID 25444548
- [Background] Kleinnijenhuis J, van Crevel R, Netea MG. Trained immunity: consequences for the heterologous effects of BCG vaccination. Trans R Soc Trop Med Hyg. 2015 Jan;109(1):29-35. doi: 10.1093/trstmh/tru168. PMID 25573107
- [Background] Higgins JP, Soares-Weiser K, Lopez-Lopez JA, Kakourou A, Chaplin K, Christensen H, Martin NK, Sterne JA, Reingold AL. Association of BCG, DTP, and measles containing vaccines with childhood mortality: systematic review. BMJ. 2016 Oct 13;355:i5170. doi: 10.1136/bmj.i5170. PMID 27737834
- [Background] Wardhana, Datau EA, Sultana A, Mandang VV, Jim E. The efficacy of Bacillus Calmette-Guerin vaccinations for the prevention of acute upper respiratory tract infection in the elderly. Acta Med Indones. 2011 Jul;43(3):185-90. PMID 21979284
- [Background] Han RF, Pan JG. Can intravesical bacillus Calmette-Guerin reduce recurrence in patients with superficial bladder cancer? A meta-analysis of randomized trials. Urology. 2006 Jun;67(6):1216-23. doi: 10.1016/j.urology.2005.12.014. PMID 16765182
- [Background] Hatherill M, Geldenhuys H, Pienaar B, Suliman S, Chheng P, Debanne SM, Hoft DF, Boom WH, Hanekom WA, Johnson JL. Safety and reactogenicity of BCG revaccination with isoniazid pretreatment in TST positive adults. Vaccine. 2014 Jun 30;32(31):3982-8. doi: 10.1016/j.vaccine.2014.04.084. Epub 2014 May 9. PMID 24814553
- [Background] Leentjens J, Kox M, Stokman R, Gerretsen J, Diavatopoulos DA, van Crevel R, Rimmelzwaan GF, Pickkers P, Netea MG. BCG Vaccination Enhances the Immunogenicity of Subsequent Influenza Vaccination in Healthy Volunteers: A Randomized, Placebo-Controlled Pilot Study. J Infect Dis. 2015 Dec 15;212(12):1930-8. doi: 10.1093/infdis/jiv332. Epub 2015 Jun 12. PMID 26071565
- [Background] Mangtani P, Abubakar I, Ariti C, Beynon R, Pimpin L, Fine PE, Rodrigues LC, Smith PG, Lipman M, Whiting PF, Sterne JA. Protection by BCG vaccine against tuberculosis: a systematic review of randomized controlled trials. Clin Infect Dis. 2014 Feb;58(4):470-80. doi: 10.1093/cid/cit790. Epub 2013 Dec 13. PMID 24336911
- [Background] Kemp EB, Belshe RB, Hoft DF. Immune responses stimulated by percutaneous and intradermal bacille Calmette-Guerin. J Infect Dis. 1996 Jul;174(1):113-9. doi: 10.1093/infdis/174.1.113. PMID 8655980
- [Background] Randomised controlled trial of single BCG, repeated BCG, or combined BCG and killed Mycobacterium leprae vaccine for prevention of leprosy and tuberculosis in Malawi. Karonga Prevention Trial Group. Lancet. 1996 Jul 6;348(9019):17-24. PMID 8691924
- [Background] To KK, Tsang OT, Leung WS, Tam AR, Wu TC, Lung DC, Yip CC, Cai JP, Chan JM, Chik TS, Lau DP, Choi CY, Chen LL, Chan WM, Chan KH, Ip JD, Ng AC, Poon RW, Luo CT, Cheng VC, Chan JF, Hung IF, Chen Z, Chen H, Yuen KY. Temporal profiles of viral load in posterior oropharyngeal saliva samples and serum antibody responses during infection by SARS-CoV-2: an observational cohort study. Lancet Infect Dis. 2020 May;20(5):565-574. doi: 10.1016/S1473-3099(20)30196-1. Epub 2020 Mar 23. PMID 32213337
- [Background] Chen Y, Li L. SARS-CoV-2: virus dynamics and host response. Lancet Infect Dis. 2020 May;20(5):515-516. doi: 10.1016/S1473-3099(20)30235-8. Epub 2020 Mar 23. No abstract available. PMID 32213336
- [Background] Giamarellos-Bourboulis EJ, Tsilika M, Moorlag S, Antonakos N, Kotsaki A, Dominguez-Andres J, Kyriazopoulou E, Gkavogianni T, Adami ME, Damoraki G, Koufargyris P, Karageorgos A, Bolanou A, Koenen H, van Crevel R, Droggiti DI, Renieris G, Papadopoulos A, Netea MG. Activate: Randomized Clinical Trial of BCG Vaccination against Infection in the Elderly. Cell. 2020 Oct 15;183(2):315-323.e9. doi: 10.1016/j.cell.2020.08.051. Epub 2020 Sep 1. PMID 32941801
- See also: Virscan — https://cdi.bio/antygen-virscan-phip-seq-service/